CLINICAL TRIAL: NCT06717594
Title: PK/PD Relationship of CAZ/AVI and FOS in the Treatment of Patients With Infections Due to Carbapenem-resistant Enterobacterales (CRE)
Brief Title: PK/PD Relationship of CAZ/AVI and FOS in the Treatment of Patients With Infections Due to CRE
Acronym: CAVIFOS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CAVIFOS; JPIAMR-ACTION (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Gram Negative Infections; Antimicrobial Resistance (AMR)
Keywords: Gram negative infection; Ceftazidime/Avibactam; Fosfomycin; Pharmacokinetics/Pharmacodynamics targets; Carbapenem-resistant Enterobacterales (CRE)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Serum samples for PK/PD analysis
  * Isolated bacterial strains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Carbapenem-resistant Enterobacterales (CRE) infection treated with CAZ/AVI ± FOS: Adult patients treated for ≥ 48 hours with CAZ/AVI or CAZ/AVI plus FOS for a microbiologically documented CRE infection

SUMMARY:
A multicenter international prospective observational pharmacological study in adult patients (≥18 years) treated with ceftazidime/avibactam (CAZ/AVI) alone or with CAZ/AVI plus fosfomycin (FOS) for infection due to carbapenem-resistant Enterobacterales (CRE) (KPC and/or OXA-48).

DETAILED DESCRIPTION:
Gram-negative infections, particularly those caused by carbapenem-resistant Enterobacterales (CRE), have a dramatic impact on patient survival. Despite the introduction of new drugs in the last years have improved the outcome of patients with CRE infections, mortality and relapse rates are still relevant, especially in patients with high-risk source as pneumonia, and those in which the attainment of optimal exposure could be reduced by underlying renal disease. The use of combination regimen in these scenarios has been proposed. However, a standardized approach is still missing. Since several in vitro studies have highlighted the synergistic effect of fosfomycin (FOS) with different antibiotic classes, including cephalosporins such drug could be an appealing option in combination therapy for the management of CRE infections.

In particular, the primary aim of the study is to assess the probability of achieving a pre-defined target of efficacy in patients treated with ceftazidime/avibactam (CAZ/AVI) and/or FOS according to different modes of drug administration in patients with CRE infections.

Secondary aim is to assess the association between plasma drug concentration of both CAZ/AVI and FOS and patient response.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the informed consent
* Age ≥ 18 years
* Adult patients treated for ≥ 48 hours with CAZ/AVI or CAZ/AVI plus FOS for a microbiologically documented CRE infection

Exclusion Criteria:

* Polymicrobial/mixed infections with exception of cases with multiple Enterobacterales susceptible to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with infection due to a difficult-to-treat Gram-negative bacteria, treated with CAZ/AVI alone or CAZ/AVI plus FOS, hospitalized during the study period in the participating centers, will be screened for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
PK/PD efficacy targets for study drugs | From enrollment (treatment onset) to 48 and 72 hours after starting treatment
  The primary endpoint will be the attainment of the pre-defined PK/PD target of efficacy at 48 and 72 hours after starting treatment for Carbapenem-resistant Enterobacterales (CRE) infection

SECONDARY OUTCOMES:
Difference in SOFA score | From day 0 (day of index positive culture) and day 7
  Difference in SOFA score between day 0 (day of treatment onset) and day 7
Trend of C-Reactive Protein (CRP) and Procalcitonin (PCT) | From day 0 (day of index positive culture) and day 7
  Trend of C-Reactive Protein (CRP) and Procalcitonin (PCT) from day 0 to day 7 after treatment onset
Microbiological eradication | From day 0 (day of index positive culture) and day 7
  Microbiological eradication defined as bacteraemia clearance or negativization of index diagnostic sample within 7 days from treatment onset
Relapse and/or reinfection | From enrollment to the end of the follow-up at three months
  Relapse (new infection with the same pathogen emerging after treatment) and/or reinfection (new infection with a different pathogen emerging after treatment) rates at day 90
All-cause mortality | From enrollment to the end of the follow-up at three months
  All-cause mortality at day 30 and at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Giannella, MD PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy
- Instituto de Biomedicina de Sevilla (IBiS), Hospital Virgen Macarena/CSIC/Universidad de Sevilla, Seville, Seville, Spain